CLINICAL TRIAL: NCT06349330
Title: The Immediate Effectiveness of a 3D Intraoral Scanner as an Adjunctive Oral Hygiene Educational Tool: A Randomized Controlled Trial
Brief Title: The Immediate Effectiveness of a 3D Intraoral Scanner as an Oral Hygiene Educational Tool
Acronym: 3D scanner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022/00908
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Periodontal Diseases; Plaque Induced Gingival Disease
Keywords: Oral hygiene instruction; Oral hygiene education
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: This is a parallel-arm randomized controlled trial and subjects are randomized into test and control groups via block randomization.
  To investigate the immediate effectiveness on the use of 3D intraoral scanner in the improvement of oral hygiene in two (2) parallel arm study with 52 subjects (n=52). The study will take place over 1 visit.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D intra-oral scanner (Experimental): Subjects will undergo 3D scanning and the 3D rendered image will be used to facilitate oral hygiene instructions.
  Interventions: Device: Test: 3D intra-oral scanner
- Standard oral hygiene (Active Comparator): Subjects will receive standard oral hygiene instructions with hand mirror.
  Interventions: Other: Control: Standard oral hygiene

INTERVENTIONS:
Device: Test: 3D intra-oral scanner — 3D intra-oral scanner will be used to scan the subjects after plaque staining is performed. Subsequently, a 3D rendered image will be produced. Participants will be given oral hygiene education and instruction before being instructed to brush.
  A cooling-off period of 30 minutes is given before participants are instructed to brush.
  Arms: 3D intra-oral scanner
Other: Control: Standard oral hygiene — Standard oral hygiene instructions will be delivered using a hand mirror. No 3D intraoral scanner will be used.
  Arms: Standard oral hygiene

SUMMARY:
The goal of this randomized controlled clinical trial is to compare the immediate effectiveness of 3D intra-oral scanners and standard oral hygiene instructions in improving the oral hygiene of 52 subjects. The main question[s] it aims to answer are:

* Does a 3D intra-oral scanner facilitate the improvement of oral hygiene in subjects?
* Does a 3D-rendered image of plaque-stained teeth confer better visualization to subjects?

Prospective Open Cohort study: Patients referred to NUCOHS Periodontology Department will be invited to participate in the study. Included participants will be randomized into the 3D scanner (test) and standard oral hygiene (control) group. Subsequently, both groups will receive personalized oral hygiene instructions before brushing their teeth. The participants will receive plaque disclosing again to compare the differences between baseline and post-intervention.

Routine periodontal parameters will be recorded at baseline and researchers will compare the percentage improvement in full mouth plaque scores to see if the test group performed better than the control group.

A questionnaire will be given to subjects in the test and control group for qualitative analysis.

The study will require 1 visit.

DETAILED DESCRIPTION:
Subjects:

The randomized controlled study will include 52 healthy volunteers from the National University Centre of Oral Health (NUCOHS), Department of Periodontology. The sample size is calculated with the assumption of a large Cohen effect size. The subjects are patients undergoing periodontal therapy in the center. After written informed consent has been obtained, the baseline periodontal parameters will be obtained to assess for inclusion and exclusion criteria. Successfully included participants will be randomized into 2 groups by blinded study team members.

There will be 2 groups:

1. Test (n=26): 3D intra-oral scanning group.
2. Control (n=26): standard oral hygiene instructions (no 3D intra-oral scanning).

Examiner:

* The blinded examiner will perform the baseline examination and the post-intervention examination.
* An unblinded examiner will perform either a) intra-oral scanning and give tailored OHI and OHE using the 3D rendered image or b) give OHI and OHE using conventional models. A standardized protocol for OHI and OHE is given to calibrate the overall instructions given.
* The standardized protocol will include a demonstration of the modified bass technique using a tooth model as well as intra-orally. Interdental brushes (Curaprox) will be fitted according to the size of the interdental gap using the Curaprox Interproximal Access Probe (IAP PROBE). Its use will be demonstrated intra-orally using a hand mirror in both groups.
* Based on the design of the study, there will be no deviation from standard periodontal treatment protocol with the exception that the test group will receive 3D intraoral scanning during oral hygiene education and instructions.
* At the end of the visit, participants from both test and control group will be given a short questionnaire by delegated study team members to evaluate their perspectives on 3D scanning (test) and standard oral hygiene (control).

Results collection:

- The delegated study member will collect the data collected during the clinical periodontal examination that has been recorded during the visit.

Primary outcome: Difference in the full mouth plaque score (%). Secondary outcomes: Participants experience/satisfaction in the test/control group on the given method of oral hygiene instruction.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy patients (ASA I and ASA II)
2. ≥ 20 teeth, excluding impacted third molars
3. , between ages 21 and 75 years
4. plaque score (PS) ≥ 50%
5. Bleeding on probing ≥ 30% of sites
6. At least 1 molar is present on each sextant
7. Probing pocket depths (PPD) should be ≤ 6 mm (h) Willingness to give consent

Exclusion Criteria:

1. Presence of PPD ≥ 7 mm, excluding the distal of 7s due to impacted wisdom teeth
2. Presence of fixed retainers
3. Presence of fixed orthodontic appliances
4. Pregnant and lactating patients
5. Cognitive impairments
6. Initiation of antibiotic therapy or antiseptic mouth rinse within 2 weeks before the study
7. Patients with known neuromotor deficits e.g. Parkinsonism, Dementia, Alzheimer's Disease
8. Diseases or medications, medications that may affect treatment
9. Heavy smokers ≥ 10 sticks/day,
10. Unwillingness to undergo periodontal treatment
11. Uncontrolled diabetes mellitus and hypertension
12. Teeth with crowns and bridges
13. Unwillingness to undergo the proposed protocol

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Full mouth plaque score (%) | Immediate/1 day
  Difference in Full Mouth Plaque Score using the two tone plaque disclosing liquid by Curaprox

SECONDARY OUTCOMES:
Patient's satisfaction of 3D scanner and standard oral hygiene group based on 5-point Likert Scale | Immediate/1 day
  Patient's acceptability to the control and intervention will be measured by a 5-point Likert scale questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Tong Lu Jacinta Dr, Principal Investigator — National University Centre for Oral Health
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doi K, Yoshiga C, Kobatake R, Kawagoe M, Wakamatsu K, Tsuga K. Use of an intraoral scanner to evaluate oral health. J Oral Sci. 2021 Jun 29;63(3):292-294. doi: 10.2334/josnusd.21-0048. Epub 2021 Jun 9. PMID 34108300
- [Background] Jung K, Giese-Kraft K, Fischer M, Schulze K, Schlueter N, Ganss C. Visualization of dental plaque with a 3D-intraoral-scanner-A tool for whole mouth planimetry. PLoS One. 2022 Oct 26;17(10):e0276686. doi: 10.1371/journal.pone.0276686. eCollection 2022. PMID 36288348